CLINICAL TRIAL: NCT01322282
Title: A Randomized, Open-Label, Single-Dose, Three-Period Crossover Bioequivalence Study to Compare an Orodispersible Tablet (ODT) Formulation of Cetirizine HCl 10 mg Taken With and Without Water Compared With a Standard Marketed 10 mg Tablet Taken With Water
Brief Title: To Test Bioequivalence Between Two Tablet Formulations in the Treatment of Allergy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: McNeil AB (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CETALY1006
Record Dates: First submitted 2011-03-23; First posted 2011-03-24 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Allergy
MeSH Terms: conditions — Hypersensitivity | interventions — Cetirizine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- ODT with Water (Experimental): Experimental Cetirizine 10 mg Orodispersible Tablet (ODT) taken with 240 mL of water
  Interventions: Drug: Cetirizine
- ODT Without Water (Experimental): Experimental Cetirizine 10 mg Orodispersible Tablet (ODT) taken without 240 mL of water
  Interventions: Drug: Cetirizine
- FCT with Water (Active Comparator): Marketed Cetirizine 10 mg Film-Coated Tablet (FCT) taken with 240 mL of water
  Interventions: Drug: Cetirizine

INTERVENTIONS:
Drug: Cetirizine — A single 10 mg dose of an experimental Cetirizine Orodispersible Tablet (ODT), with a 7-day washout period between visits
  Other Names: Not yet marketed
  Arms: ODT Without Water; ODT with Water
Drug: Cetirizine — A single 10 mg dose of a marketed Cetirizine Film-Coated Tablet (FCT), with a 7-day washout period between visits
  Other Names: Benadryl One A Day 10 mg Film-Coated Tablet
  Arms: FCT with Water

SUMMARY:
This study is designed to assess bioequivalence between two products used for treatment of allergy.

DETAILED DESCRIPTION:
This study is designed to evaluate if a test formulation of cetirizine 10 mg orodispersible tablet (ODT) taken with and without water is bioequivalent to a marketed reference formulation of cetirizine 10 mg tablet (Benadryl One A Day, McNeil Products Ltd, UK) taken with water. This study will also evaluate the tolerability of test and reference formulations.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects
* Volunteers aged of at least 18 years but not older than 55 years
* Subjects will have a Body Mass Index (BMI) greater than or equal to 18.50 and below 30.00 kg/m2
* Non- or ex-smokers; an ex-smoker being defined as someone who completely stopped smoking for at least 12 months before day 1 of this study
* Clinical laboratory values within the laboratory's stated normal range; if not within this range, they must be without any clinical significance
* Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on physical examination and/or clinical laboratory evaluations (hematology, biochemistry, ECG and urinalysis)
* Has signed and dated the informed consent document, indicating that the subject has been informed of all pertinent aspects of the study
* Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion Criteria:

* Seated pulse rate below 45 bpm or higher than 90 bpm at screening
* Seated blood pressure below 90/60 mmHg or higher than 140/90 mmHg at screening
* Relationship to persons involved directly with the conduct of the study (i.e., principal investigator; sub-investigators; study coordinators; other study personnel; employees or contractors of the sponsor or Johnson & Johnson subsidiaries; and the families of each)
* Presence of any tongue piercings
* Presence of braces
* Females who are pregnant or are lactating
* Females of childbearing potential or males with a female partner of childbearing potential who refuse to use an acceptable contraceptive regimen throughout the entire duration of the study
* Females who are pregnant according to a positive serum pregnancy test
* Any medical history or condition, or use of any drug or medication, that the investigator determines could compromise subject safety or the evaluation of results.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration | During 32 hours post-dose
  Maximum Observed Plasma Concentration (Cmax), which is the maximum (peak) concentration (amount of drug) measurable in blood plasma after a dose is administered, measured in nanograms/milliliter (ng/mL)
Bioavailability [AUC(0-t)] | During 32 hours post-dose
  Bioavailability [AUC(0-t)] is a measure of how much of the drug reaches the person's bloodstream within a given period of time for the body to use. The extent of product bioavailability is estimated by the area under the blood concentration vs time curve. The Area Under the Curve (AUC) is calculated by plotting the drug's blood levels on a graph at different times during the set period. The area under this curve reflects the amount of drug exposure in the set time period, calculated as hour * nanograms (ng) per milliliter (mL).
Bioavailability Extrapolated to Infinity [AUC (0-∞)] | 32 hours post-dose
  Bioavailability Extrapolated to Infinity [AUC (0-∞)] is a calculated measure of how much of the drug will ever reach the person's bloodstream for the body to use. AUC (0-∞) stands for the area under the plasma concentration versus time curve from time zero (pre-dose) to extrapolated infinite time (forever). It is obtained from calculating AUC (0-t) plus AUC (t-∞).

SECONDARY OUTCOMES:
Time of Maximum Concentration | During 32 hours post-dose
  The time at which maximum concentration is reached (Tmax)
Terminal Elimination Rate Constant | During 32 hours post-dose
  The Terminal Elimination Rate Constant (Lamda z) is the time required to eliminate half the administered dose
Terminal Phase Plasma Half-Life | During 32 hours post-dose
  Terminal phase plasma half-life (t ½) is the time required to divide the plasma concentration by two after reaching pseudo-equilibrium, rather than the time required to eliminate half the administered dose.
Area under the Curve to the Tmax of the Reference Products | During 32 hours post-dose
  Area under the plasma concentration versus time curve to the time of the maximum concentration of the reference products (AUCReftmax)
Relative percentage of AUCT with respect to AUC∞ (AUCT/∞) | During 32 hours post-dose
  AUCT is the area under the plasma concentration verses time curve from start of drug administration until the time of the last measurable plasma concentration.
  AUC∞ is the area under the plasma concentration versus time curve from start of drug administration until extrapolated infinite time.
  AUCT/ AUC∞ is an inversed measure of how large the extrapolated area under the curve is.
Mean Residence Time | During 32 hours post-dose
  The average amount of time a particle (e.g., a drug substance molecule) remains in a compartment or system.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Kruse, PhD, Study Director — McNeil AB
Locations (1):
- Algorithme Pharma Inc., Mount Royal, Quebec, Canada